CLINICAL TRIAL: NCT04448548
Title: Possible Roles of MDW in Infection Management in Emergency Care
Status: Completed | Type: Observational
Sponsor: Szeged University (Other)
Responsible Party: Sponsor
Other Study IDs: MDW
Record Dates: First submitted 2020-06-24; First posted 2020-06-26 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Infection; Sepsis
MeSH Terms: conditions — Infections; Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: blood sample taking — For study purposes, blood sample was taken during the first medical examination from patients with suspected infection.

SUMMARY:
A retrospective study to determine the potential value of MDW among other biomarkers in the diagnosis of infection.

DETAILED DESCRIPTION:
MDW as a novel indicator can be useful in clinical practice in the emergency care. However, until now, no study has been published about MDW's general relationship and coherence with multiple, conventional laboratory tests for infections, such as PCT, C-reactive protein (CRP), WBC, neutrophil count (NC), neutrophil percentage and immature granulocyte count (IGC) together.

ELIGIBILITY:
Inclusion Criteria:

* adult (18+ years), receiving care for suspected infection

Exclusion Criteria:

* refuses to sign the consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult (18+ years), receiving care for suspected infection
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
MDW cutoff value for infection | 4 months
  Cutoff value for MDW indicating infection

CONTACTS AND LOCATIONS:
Locations (1):
- University of Szeged, Emergency Department, Szeged, Hungary